CLINICAL TRIAL: NCT06447623
Title: Study of Efficacy of Apatinib Combined With cdk4/6i in First-line Treatment for HR+/HER2- SNF4 Subtype Advanced Breast Cancer (Open, Randomized, Phase III)
Brief Title: Apatinib Combined With cdk4/6i in First-line Treatment for HR+/HER2- SNF4 Subtype Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N068
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Advanced Breast Cancer; HR+/HER2- Breast Cancer
Keywords: HR+/HER2- breast cancer; Advanced Breast Cancer
MeSH Terms: interventions — apatinib; Aromatase Inhibitors; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm-A (Experimental): Apatinib combined with cdk4/6i and Endocrine therapy.
  Interventions: Drug: Apatinib; Drug: CDK4/6 Inhibitor; Drug: Aromatase inhibitor and Fulvestrant
- Arm-B (Active Comparator): cdk4/6i and Endocrine therapy.
  Interventions: Drug: CDK4/6 Inhibitor; Drug: Aromatase inhibitor and Fulvestrant

INTERVENTIONS:
Drug: Apatinib — Apatinib is a kind of TKI inhibitor.
  Arms: Arm-A
Drug: CDK4/6 Inhibitor — Dalpiciclib (SHR6390) is a kind of CDK4/6 inhibitor that has demonstrated tolerability and preliminary clinical activity in patients with heavily pretreated hormone receptor-positive, HER2-negative advanced breast cancer.
Drug: Aromatase inhibitor and Fulvestrant — Endocrine therapy combined with CDK4/6 inhibitors is the standard first-line therapy for advanced luminal breast cancer. Investigators choose endocrine therapy including Letrozole, Anastrozole, Exemestane, and Fulvestrant. Postmenopausal participants should use Goserelin.

SUMMARY:
This is a randomized, controlled, open-label, phase III study to explore the efficacy and safety of Apatinib in combination with standard first-line endocrine therapy for the HR+/ HER2-SNF4 subtype of advanced breast cancer. The study was used to explore the efficacy of Apatinib in combination with standard endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Patients need to meet all of the following conditions

  * Patients must be ≥18 and ≤ 75 years of age;
  * Pathologically confirmed breast cancer is HR+/HER2- breast cancer (IHC ER >10%, or/and PR>10%, HER 0 OR +, if HER2++, FISH negative);
  * SNF4 subtype definition: SNF4 subtype confirmed by digital pathology of H&E sections;
  * Locally advanced breast cancer (radical local therapy is not possible) or metastatic breast cancer (without using adjuvant CDK4/6 inhibitors in the past, or one year after adjuvant CDK4/6 inhibitor therapy has ended);
  * No prior therapy (chemotherapy, targeted therapy, etc.) for advanced or metastatic breast cancer;
  * Patients with at least one measurable lesion that has not previously received radiation therapy and can be evaluated repeatedly according to RECIST 1.1;
  * The functions of the main organs are basically normal, and the following conditions are met:

    1. Blood routine examination standards should meet: HB≥90g/L (no blood transfusion within 14 days); ANC≥1.5×109/L; PLT≥75×109/L;
    2. Biochemical examination shall meet the following standards: TBIL≤1.5×ULN (upper limit of normal value); ALT and AST≤3 x ULN; In case of liver metastasis, ALT and AST≤5×ULN; Serum Cr ≤1.5×ULN, endogenous creatinine clearance > 50ml/min (Cockcroft-Gault formula);
  * ECOG performance status 0 or 1; The expected survival is more than 3 months;
  * Fertile female is required to use a medically approved contraceptive during study treatment and for at least 3 months after the last use of the study drug;
  * Patients voluntarily join the study, sign the informed consent, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

* Patients with any of the following conditions were excluded from the study

  * Patients with central nervous system metastasis out of control (symptoms need to use glucocorticoids or mannitol).
  * A history of clinically significant or uncontrolled heart disease, including congestive heart failure, angina pectoris, myocardial infarction within the last 6 months, or ventricular arrhythmia;
  * Radiotherapy, chemotherapy, surgery, other targeted therapy, and immunotherapy for advanced HR+/HER2- breast cancer within 4 weeks before the first administration of drugs used in this study.
  * Pregnant or lactating patients;
  * Other malignancies within the previous 3 years, excluding cured skin basal cell carcinoma and cervical carcinoma in situ;
  * Significant comorbid medical conditions, including mental illnesses that the investigator or sponsor believes would adversely affect the patient's participation in the study;
  * Allergic physique, or known allergic history of the drug components of this program; Or allergic to other monoclonal antibodies;
  * The investigator does not consider the patient suitable for participation in any other circumstances of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Approximately 5 years
  The interval from randomization until the first occurrence of disease progression (according to RECIST 1.1) or death from any cause, which ever occurs first.

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) | Approximately 5 years
  CBR is the total percentage of participants who achieved a complete response, partial response, or had stable disease for 6 months or more.
Objective Response Rate (ORR) | Approximately 5 years
  ORR is defined as the proportion of participants who have a complete response (CR) or partial response (PR) based on BICR and investigator assessment using RECIST 1.1.
Overall Survival (OS) | Approximately 5 years
  OS is defined as the time from randomisation until the date of death due to any cause.
Safety and tolerability | Approximately 5 years
  Number of adverse events according to NCI-CTCAE Version 5.0 per each treatment arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No